CLINICAL TRIAL: NCT02403219
Title: Paralysis of the Orbicularis Muscle of the Eye by Using Botulinum Toxin Type A in the Treatment for Dry Eye
Brief Title: Paralysis of the Orbicularis Muscle of the Eye in the Treatment for Dry Eye
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CEI-2013-/06/06
Record Dates: First submitted 2015-01-21; First posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Dry Eye Syndromes
Keywords: Dry eye; Botulinum toxin A; Orbicularis muscle of the eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botulinum toxin type A injection (Experimental): An injection of 4 international units of botulinum toxin type A will be applied in the medial in the medial part of the lower eyelid near the punctum directed along the medial canthal tendon in a single application by subcutaneous injection.
  Interventions: Drug: Botulinum toxin type A injection
- Sham injection (Sham Comparator): An injection of 4 international units of sham will be applied in the medial in the medial part of the lower eyelid near the punctum directed along the medial canthal tendon in a single application by subcutaneous injection.
  Interventions: Other: Saline solution injection

INTERVENTIONS:
Drug: Botulinum toxin type A injection — Injection of botulinum toxin type A
  Other Names: Botox
  Arms: Botulinum toxin type A injection
Other: Saline solution injection — Injection of saline solution
  Other Names: Saline solution
  Arms: Sham injection

SUMMARY:
This is a prospective, comparative, contralateral eye study. Patients older than 18 years who have had treatment with topical lubricants for at least 1 month and persist with symptoms of dry eye and corneal staining with fluorescein were included. Patients with dry eye attributable to abnormalities of the eyelids, nasolacrimal obstruction and active corneal infection, as well as patients with severe dry eye were excluded from the study. One eye randomly received a subcutaneous injection of botulinum toxin in the medial part of the lower eyelid, and the other eye received a similar procedure with placebo. The subjective evaluation was achieved with a questionnaire assessing symptoms of dry eye and conjunctivitis, quality of vision and ocular comfort level each eye separately. The objective evaluation included the measurement of the tear film break up time, Schirmer's test and with a modification of the Oxford grading scheme for corneal and conjunctival staining.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with topical lubricants for at least 1 month and persist with symptoms of dry eye and corneal staining with fluorescein.

Exclusion Criteria:

* Dry eye patients attributable to abnormalities of the eyelids (problems with the mechanism of blinking, poor eyelid position, changes in position or structure of the eyelashes, high surface lesions, etc.)
* Nasolacrimal obstruction.
* Active corneal infection.
* Patients with severe grade 4 dry eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2014-02 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Symptoms of dry eye (questionnaire) | 6 months
  A questionnaire assessing symptoms of dry eye each eye separately, including dryness, watery eyes, itching, burning, foreign body, fluctuating vision and light sensitivity. Depending on the frequency, each symptom will be graded from 0 to 5.
Symptoms of conjunctivitis (questionnaire) | 6 months
  A questionnaire assessing symptoms of conjunctivitis eye separately, including redness and discharge. Depending on the frequency, each symptom will be graded from 0 to 5.
Quality of vision (graded perception of patient) | 6 months
  The quality of vision will be graded from 0 to 5 according to the perception of the patient.
Ocular comfort level (graded perception of patient) | 6 months
  The ocular comfort level will be graded from 0 to 5 according to the perception of the patient.
Moisturizing agent usage (patient will be asked how many times a day does he use the moisturizing agent and will be graded from 0 to 5 according to the frequency) | 6 months
  The
Visual acuity (Snellen vision acuity) | 6 months
  Snellen vision acuity
Measurement of the tear film break up time (After fluorescein staining, the time required for dry spots to appear on the corneal surface after blinking) | 6 months
  After fluorescein staining, the time required for dry spots to appear on the corneal surface after blinking will be recorded in seconds.
Schirmer's test | 6 months
  After instillation of topical anesthetic, paper strips are inserted into the conjunctival sac for 5 minutes to measure the production of tears in millimeters.
Oxford grading scheme for corneal and conjunctival staining | 6 months
  After fluorescein staining, the corneal and conjunctival staining will be graded according to severity from 0 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Serna-Ojeda, MD, Principal Investigator — Instituto de Oftalmologia Conde de Valenciana; Ángel Nava-Castañeda, MD, Study Director — Instituto de Oftalmologia Conde de Valenciana

REFERENCES:
- [Background] The definition and classification of dry eye disease: report of the Definition and Classification Subcommittee of the International Dry Eye WorkShop (2007). Ocul Surf. 2007 Apr;5(2):75-92. doi: 10.1016/s1542-0124(12)70081-2. PMID 17508116
- [Background] Horwath-Winter J, Bergloeff J, Floegel I, Haller-Schober EM, Schmut O. Botulinum toxin A treatment in patients suffering from blepharospasm and dry eye. Br J Ophthalmol. 2003 Jan;87(1):54-6. doi: 10.1136/bjo.87.1.54. PMID 12488263
- [Background] Sahlin S, Chen E, Kaugesaar T, Almqvist H, Kjellberg K, Lennerstrand G. Effect of eyelid botulinum toxin injection on lacrimal drainage. Am J Ophthalmol. 2000 Apr;129(4):481-6. doi: 10.1016/s0002-9394(99)00408-0. PMID 10764857
- [Background] Reifler DM. Early descriptions of Horner's muscle and the lacrimal pump. Surv Ophthalmol. 1996 Sep-Oct;41(2):127-34. doi: 10.1016/s0039-6257(96)80002-6. PMID 8890438
- [Background] Kakizaki H, Zako M, Miyaishi O, Nakano T, Asamoto K, Iwaki M. The lacrimal canaliculus and sac bordered by the Horner's muscle form the functional lacrimal drainage system. Ophthalmology. 2005 Apr;112(4):710-6. doi: 10.1016/j.ophtha.2004.11.043. PMID 15808266